CLINICAL TRIAL: NCT03771755
Title: A Prospective, Randomized, Double-blind Study Assessing the Efficacy of Intravenous (IV) Ibuprofen Versus IV Acetaminophen for the Treatment of Pain Following Orthopaedic Low Extremity Surgery
Brief Title: Ibuprofen IV vs Acetaminophen IV for the Treatment of Pain Following Orthopaedic Low Extremity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes026
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Lower Extremity Problem; Surgery; Postoperative Pain
Keywords: ibuprofen; acetaminophen; orthopedic; VAS; morphine; opioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen group (Active Comparator): 800 mg IV - Ibuprofen every 6 hours. In case required - followed with Morphine (PCA) 1-2 mg every 5 minutes
  Interventions: Drug: Ibuprofen
- Acetaminophen group (Placebo Comparator): 1000mg IV Acetaminophen every 6 hours. In case required - followed with Morphine (PCA) 1-2 mg every 5 minutes
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — 800 mg IV - Ibuprofen every 6 hours. In case required - followed with Morphine (PCA) 1-2 mg every 5 minutes
  Arms: Ibuprofen group
Drug: Acetaminophen — 1000mg IV Acetaminophen every 6 hours. In case required - followed with Morphine (PCA) 1-2 mg every 5 minutes
  Arms: Acetaminophen group

SUMMARY:
This study aims to evaluate the efficacy of IV Ibuprofen versus IV Acetaminophen in the reduction of pain following orthopedic low extremity procedures

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Patients undergoing orthopedic low extremity surgery were screened. Eligible subjects were then randomized into treatment group (intravenous ibuprofen) and control group (intravenous acetaminophen). In case required, patients from both group will be given Morphine (PCA) 1-2 mg every 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Orthopedic Low Extremity Surgery with general anesthesia and anticipated need post operative IV analgesia with anticipated use of >48 hours.
* Adequate IV access.
* Anticipated hospital stay>48 hours.
* Age 18-70 years old with physical status ASA I- III.
* Patients able to fill informed consent sheet.

Exclusion Criteria:

* patients with use of analgesia, muscle relaxants, NSAIDs and sedatives less than 24 hours to study drug administration
* anemia (active, clinically significant anemia) and/or a history or evidence of asthma or heart failure
* historical or at higher risk intracerebral bleeding, history of allergy or hypersensitive to NSAID, Ibuprofen, Acetaminophen or opioid
* pregnant or nursing
* body weight less than 30 kg
* any active clinically significant bleeding or have underlying platelet dysfunction and/or receiving full dose anticoagulation therapy
* GI bleeding that required medical intervention within the previous 6 weeks (unless definitive surgery has been performed)
* on dialysis or renal dysfunction
* impaired liver function
* inability to achieve hemostasis or inability to close surgical incision prior to operating room discharge
* operative procedure includes organ transplant, pre-and intra- operative procedure utilized for the prevention of pre- or post-operative pain (i.e, epidural or nerve blocks)
* received anoher investigational drug within the past 30 days
* known or suspected history of alcohol or drug abuse
* severe infection and/or inflammatory disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 24 hours
  demonstrated by the measurement VAS (Visual Analog Scale) for 24 hrs postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Kehlet H, Holte K. Effect of postoperative analgesia on surgical outcome. Br J Anaesth. 2001 Jul;87(1):62-72. doi: 10.1093/bja/87.1.62. No abstract available. PMID 11460814
- [Background] Shavit Y, Fridel K, Beilin B. Postoperative pain management and proinflammatory cytokines: animal and human studies. J Neuroimmune Pharmacol. 2006 Dec;1(4):443-51. doi: 10.1007/s11481-006-9043-1. Epub 2006 Sep 29. PMID 18040817
- [Background] Beilin B, Shavit Y, Trabekin E, Mordashev B, Mayburd E, Zeidel A, Bessler H. The effects of postoperative pain management on immune response to surgery. Anesth Analg. 2003 Sep;97(3):822-827. doi: 10.1213/01.ANE.0000078586.82810.3B. PMID 12933409
- [Background] Hall GM, Peerbhoy D, Shenkin A, Parker CJ, Salmon P. Relationship of the functional recovery after hip arthroplasty to the neuroendocrine and inflammatory responses. Br J Anaesth. 2001 Oct;87(4):537-42. doi: 10.1093/bja/87.4.537. PMID 11878721
- [Background] Esme H, Kesli R, Apiliogullari B, Duran FM, Yoldas B. Effects of flurbiprofen on CRP, TNF-alpha, IL-6, and postoperative pain of thoracotomy. Int J Med Sci. 2011 Mar 10;8(3):216-21. doi: 10.7150/ijms.8.216. PMID 21448308
- [Background] Dionne RA, Gordon SM, Rowan J, Kent A, Brahim JS. Dexamethasone suppresses peripheral prostanoid levels without analgesia in a clinical model of acute inflammation. J Oral Maxillofac Surg. 2003 Sep;61(9):997-1003. doi: 10.1016/s0278-2391(03)00310-0. PMID 12966473
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Duggan ST, Scott LJ. Intravenous paracetamol (acetaminophen). Drugs. 2009;69(1):101-13. doi: 10.2165/00003495-200969010-00007. PMID 19192939
- [Background] Glenn EM, Bowman BJ, Rohloff NA. Anti-inflammatory and PG inhibitory effects of phenacetin and acetaminophen. Agents Actions. 1977 Dec;7(5-6):513-6. doi: 10.1007/BF02111123. PMID 414527
- [Background] Vinegar R, Truax JF, Selph JL. Quantitative comparison of the analgesic and anti-inflammatory activities of aspirin, phenacetin and acetaminophen in rodents. Eur J Pharmacol. 1976 May;37(1):23-30. doi: 10.1016/0014-2999(76)90004-2. PMID 1278245
- [Background] Wolfe F, Zhao S, Lane N. Preference for nonsteroidal antiinflammatory drugs over acetaminophen by rheumatic disease patients: a survey of 1,799 patients with osteoarthritis, rheumatoid arthritis, and fibromyalgia. Arthritis Rheum. 2000 Feb;43(2):378-85. doi: 10.1002/1529-0131(200002)43:23.0.CO;2-2. PMID 10693878
- [Background] Bradley JD, Brandt KD, Katz BP, Kalasinski LA, Ryan SI. Comparison of an antiinflammatory dose of ibuprofen, an analgesic dose of ibuprofen, and acetaminophen in the treatment of patients with osteoarthritis of the knee. N Engl J Med. 1991 Jul 11;325(2):87-91. doi: 10.1056/NEJM199107113250203. PMID 2052056
- [Background] Bonnefont J, Courade JP, Alloui A, Eschalier A. [Antinociceptive mechanism of action of paracetamol]. Drugs. 2003;63 Spec No 2:1-4. French. PMID 14758785
- [Background] Graham GG, Scott KF. Mechanism of action of paracetamol. Am J Ther. 2005 Jan-Feb;12(1):46-55. doi: 10.1097/00045391-200501000-00008. PMID 15662292
- [Background] Khan AA, Iadarola M, Yang HY, Dionne RA. Expression of COX-1 and COX-2 in a clinical model of acute inflammation. J Pain. 2007 Apr;8(4):349-54. doi: 10.1016/j.jpain.2006.10.004. Epub 2007 Jan 30. PMID 17270500
- [Background] Kashefi P, Honarmand A, Safavi M. Effects of preemptive analgesia with celecoxib or acetaminophen on postoperative pain relief following lower extremity orthopedic surgery. Adv Biomed Res. 2012;1:66. doi: 10.4103/2277-9175.100197. Epub 2012 Aug 28. PMID 23459777
- [Background] Crofford LJ. Use of NSAIDs in treating patients with arthritis. Arthritis Res Ther. 2013;15 Suppl 3(Suppl 3):S2. doi: 10.1186/ar4174. Epub 2013 Jul 24. PMID 24267197
- [Background] Morris PE, Promes JT, Guntupalli KK, Wright PE, Arons MM. A multi-center, randomized, double-blind, parallel, placebo-controlled trial to evaluate the efficacy, safety, and pharmacokinetics of intravenous ibuprofen for the treatment of fever in critically ill and non-critically ill adults. Crit Care. 2010;14(3):R125. doi: 10.1186/cc9089. Epub 2010 Jun 30. PMID 20591173
- [Background] Scott LJ. Intravenous ibuprofen: in adults for pain and fever. Drugs. 2012 May 28;72(8):1099-109. doi: 10.2165/11209470-000000000-00000. PMID 22621696
- [Background] Southworth S, Peters J, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen 400 and 800 mg every 6 hours in the management of postoperative pain. Clin Ther. 2009 Sep;31(9):1922-35. doi: 10.1016/j.clinthera.2009.08.026. PMID 19843482
- [Background] Kroll PB, Meadows L, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen (i.v.-ibuprofen) in the management of postoperative pain following abdominal hysterectomy. Pain Pract. 2011 Jan-Feb;11(1):23-32. doi: 10.1111/j.1533-2500.2010.00402.x. PMID 20642488
- [Background] Singla N, Rock A, Pavliv L. A multi-center, randomized, double-blind placebo-controlled trial of intravenous-ibuprofen (IV-ibuprofen) for treatment of pain in post-operative orthopedic adult patients. Pain Med. 2010 Aug;11(8):1284-93. doi: 10.1111/j.1526-4637.2010.00896.x. Epub 2010 Jun 30. PMID 20609131
- [Background] Southworth SR, Woodward EJ, Peng A, Rock AD. An integrated safety analysis of intravenous ibuprofen (Caldolor((R))) in adults. J Pain Res. 2015 Oct 23;8:753-65. doi: 10.2147/JPR.S93547. eCollection 2015. PMID 26604816